CLINICAL TRIAL: NCT04639882
Title: Motivating Recruitment and Efficacy in Normative Feedback Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Clayton Neighbors, Professor, University of Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R21AA022369 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Heavy Drinking

STUDY DESIGN:
Intervention Model Description: Heavy drinking college students (N=498) participated in a 2 (in-person vs. remote delivery) × 2 (compensation vs. no compensation) × 2 (PNF vs. control) design with follow-up assessments occurring remotely three and six months later.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control-Remote-$0 (Experimental): In this condition, Participants:
  * receive attention control feedback
  * complete the baseline and intervention procedure remotely
  * are compensated $0 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- Control-Remote-$30 (Experimental): In this condition, Participants:
  * receive attention control feedback
  * complete the baseline and intervention procedure remotely
  * are compensated $30 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- Control-InPerson-$0 (Experimental): In this condition, Participants:
  * receive attention control feedback
  * complete the baseline and intervention procedure in the research lab
  * are compensated $0 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- Control-InPerson-$30 (Experimental): In this condition, Participants:
  * receive attention control feedback
  * complete the baseline and intervention procedure in the research lab
  * are compensated $30 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- PNF-Remote-$0 (Experimental): In this condition, Participants:
  * receive personalized normative feedback
  * complete the baseline and intervention procedure remotely
  * are compensated $0 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- PNF-Remote-$30 (Experimental): In this condition, Participants:
  * receive personalized normative feedback
  * complete the baseline and intervention procedure remotely
  * are compensated $30 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- PNF-Inperson-$0 (Experimental): In this condition, Participants:
  * receive personalized normative feedback
  * complete the baseline and intervention procedure in the research lab
  * are compensated $0 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback
- PNF-Inperson-$30 (Experimental): In this condition, Participants:
  * receive personalized normative feedback
  * complete the baseline and intervention procedure in the research lab
  * are compensated $30 for completing the baseline and intervention procedure
  Interventions: Behavioral: Personalized normative feedback

INTERVENTIONS:
Behavioral: Personalized normative feedback — Information presenting perceived and actual drinking norms.

SUMMARY:
Excessive alcohol consumption among college students continues to be a serious public health concern associated with a wide range of negative consequences. Brief computer-based social norms interventions, including personalized normative feedback (PNF), have shown consistent effects in reducing problematic drinking in this population, and there is some evidence that in-lab computer-delivered interventions may be more effective than remote interventions. Most studies have been conducted using generous incentives which may reduce the feasibility of dissemination on a larger scale and may undermine trial efficacy. In accordance with NIAAA aims, this research aims to (a) investigate delivery modality (i.e., in lab versus remotely) and incentives as important factors affecting the efficacy of PNF interventions and (b) develop intervention strategies that facilitate wider dissemination of inexpensive empirically-supported brief interventions for college students, thereby reducing problem drinking during a high-risk time period.

DETAILED DESCRIPTION:
The current application evaluates motivational factors associated with recruitment into and efficacy of brief computer-delivered interventions for heavy drinking college students. College students are at increased risk for alcohol misuse compared to other adults, and development of efficacious intervention approaches is an urgent priority for NIAAA. Over the past several years empirical evidence has demonstrated support for computer-based personalized normative feedback (PNF) interventions which correct normative misperceptions of drinking and thereby reduce drinking behavior. Two specific questions which have remained largely unaddressed include whether the effectiveness of computer-based interventions depends on the location in which they are completed, and what is the optimal incentive structure to balance recruitment with motivational biases in intervention trials. A preliminary comparison of findings across several studies suggests that remote PNF interventions may be less effective than in-lab PNF interventions. However, the evidence is not conclusive because no study provides a direct comparison between delivery methods based on random assignment within the same study. This R21 recruited 498 heavy drinking college students and randomly assigned them to a 2 × 2 × 2 repeated measures design. Participants were randomly assigned to in-lab PNF, remote PNF, in-lab attention control, or remote attention control. Participants were also randomly assigned to receive no incentive ($0) or an incentive ($30) for participation. Assessments included baseline, postintervention, 3-month, and 6-month follow-ups. College students' motivational orientations, incentives, and typical drinking are expected to moderate differences between delivery methods. We expect that students who receive incentives for participating in intervention studies will be more likely to participate, but less likely to reduce drinking because they will be more likely to attribute their participation to extrinsic motivation. Further, students who receive computer-based PNF in the laboratory for no incentive are expected to exhibit the largest reductions in drinking. In contrast, students administered attention-control feedback remotely for an incentive ($30) are expected to exhibit the smallest reductions in drinking. Perceived value of intervention, retention of intervention content, and attribution for participation are expected to mediate incentive effects and differential efficacy of in-lab versus remote delivery. This research is expected to yield theoretical and practical improvements to feedback-based intervention strategies with potential to reduce drinking and related negative consequences with a stronger theoretical basis and at lower cost than have been previously available.

ELIGIBILITY:
Inclusion Criteria:

Reporting one or more heavy drinking occasions (4/5 drinks on one drinking occasion for women/men) in the previous month Reporting one or more negative alcohol-related consequence in the previous month Being between 18 and 26 years of age Being a registered University of Houston student Providing consent to participate in the study

Exclusion Criteria:

Not meeting any of the inclusion criteria Unwillingness to participate Failure to provide consent

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 498 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of drinks in past month - Timeline Follow-back (TLFB) | 1 month
  This measure asks participants to indicate how many drinks they consumed on each day of the previous month. Scores are summed.
Number of drinks on a typical week - Daily Drinking Questionnaire (DDQ) | 3 months
  Participants are asked how many drinks they typically drink on each day of a typical week. These values are summed to create a drinks per week score. From Collins, Parks, and Marlatt (1985).
Number of peak drinks consumed | One month
  Participants are asked to indicate the maximum number of drinks consumed on one occasion.
Alcohol-related consequences: Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) | One month
  A measure of 27 alcohol consequences. Participants indicate whether they have experienced the consequence or not and responses are summed to create a total score.
Alcohol-related consequences: Rutgers Alcohol Problems Index (RAPI) | 3 months
  A measure of alcohol consequences. Participants indicate the frequency with which they have experienced each consequence; responses are summed to create a total score.

SECONDARY OUTCOMES:
Perception of number of drinks a typical college student drinks | 3 months
  The DDQ (Outcome 2) was modified to ask participants how often they think the typical college student of their same sex drinks in a typical week. Responses are again summed to create a total score. This measure is posited as a mediator of intervention efficacy on changes in drinking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No